CLINICAL TRIAL: NCT04595838
Title: A Randomized, Prospective, Multi-center Trial to Assess the Efficacy of a Cryotherapy Device Versus Best Supportive Oral Care in Mitigating Symptoms of Oral Mucositis in Patients Receiving Chemotherapy for the Treatment of Cancer
Brief Title: A Trial Assessing Chemo Mouthpiece Device With Best Supportive Care for Symptoms of Chemotherapy-Induced Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chemo Mouthpiece (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHEM-01
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Oral Mucositis
Keywords: Prospective Studies, Stomatitis, Cryotherapy, Patient Reported Outcome Measures
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm A:Best supportive oral care and Chemo Mouthpiece (Experimental): Patients will receive best supportive oral care along with using the Chemo Mouthpiece device.
  Interventions: Device: Chemo Mouthpiece
- Arm B Best supportive oral care only (Other): Patients will receive best supportive oral care only.
  Interventions: Other: Best Supportive Care only

INTERVENTIONS:
Device: Chemo Mouthpiece — Frozen tube that fills the oral cavity used during and after chemotherapy to ease and prevent symptoms of oral mucositis
  Other Names: Oral cryotherapy delivery device
  Arms: Arm A:Best supportive oral care and Chemo Mouthpiece
Other: Best Supportive Care only — Standard Oral care for Chemotherapy
  Arms: Arm B Best supportive oral care only

SUMMARY:
This study will compare the use of the Chemo MouthpieceTM device along with best supportive oral care to best supportive oral care alone to rate the effectiveness of Chemo MouthpieceTM in lessening symptoms associated with chemotherapy regimen known to place patients at risk for symptomatic mucositis and, of those, chemotherapy regimens for which ice-based cryotherapy has been demonstrated to have a favorable impact on oral mucositis symptom management. Subjects who are receiving standard chemotherapy regimens will be randomly assigned to receive either study device and oral care ingredients or oral care ingredients only. All subjects will complete daily diaries for the first 14 days of chemotherapy Cycles 1 and 2. Subjects who are assigned to the study device arm will use the device during their chemotherapy infusion in clinic and will continue to use the device at home ,at least twice daily, for the first six (6) days of chemotherapy Cycles 1 and 2. Prior to the first chemotherapy infusion in Cycle 3, all subjects in the study regardless of treatment assignment will have the option of using the Chemo MouthpieceTM for subsequent cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years
2. Planned to receive at least 2 cycles of infused stomatotoxic chemotherapy regimens such as:

   * CMF (cyclophosphamide (Cytoxan), methotrexate, 5-FU)
   * Standard AC+T regimen (doxorubicin (Adriamycin), cyclophosphamide (Cytoxan), Taxane [paclitaxel (Taxol) or docetaxel (Taxotere)]) or any combination of two or more components (e.g., ACT, TAC, TA, AT, AC)
   * ABVD (doxorubicin (Adriamycin), bleomycin, vinblastine, dacarbazine)
   * FOLFIRI (irinotecan, 5-FU, leucovorin)
   * Any other 5-FU-based regimen (excluding FOLFOX)
3. Be willing and able to complete all study-related activities
4. Properly obtained written informed consent

Exclusion Criteria:

1. Receiving any oxaliplatin-containing chemotherapy regimen, such as FOLFOX
2. Concurrent radiotherapy
3. Unable or unwilling to complete study assessments
4. Unable or unwilling to avoid using ice chips
5. Known allergy to silicone
6. Concurrent participation in another interventional clinical study or use of another investigational agent within 30 days prior to randomization
7. Any other clinical or psychiatric condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the protocol
8. Chronic use of opioid analgesics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
The incidence of oral mucositis symptomatic events observed during the first cycle of chemotherapy. | Cycle 1 of chemotherapy (14-28 days, time frame varies based on regimen)
  The presence and severity of oral mucositis symptoms will be measured by patient self-report using the Oral Mucositis Symptom Assessment scale with positive symptoms defined as a score of 1 or greater and severe symptoms defined as a score of 2 or greater.
The incidence of oral mucositis symptomatic events observed during the second cycle of chemotherapy. | Cycle 2 of chemotherapy (14-28 days, time frame varies based on regimen)
  The presence and severity of oral mucositis symptoms will be measured by patient self-report using the Oral Mucositis Symptom Assessment scale with positive symptoms defined as a score of 1 or greater and severe symptoms defined as a score of 2 or greater.
The incidence of severe oral mucositis symptomatic events observed during the first cycle of chemotherapy. | Cycle 1 of chemotherapy (14-28 days, time frame varies based on regimen)
  The presence and severity of oral mucositis symptoms will be measured by patient self-report using the Oral Mucositis Symptom Assessment scale with positive symptoms defined as a score of 1 or greater and severe symptoms defined as a score of 2 or greater.
The incidence of severe oral mucositis symptomatic events observed during the second cycle of chemotherapy. | Cycle 2 of chemotherapy (14-28 days, time frame varies based on regimen)
  The presence and severity of oral mucositis symptoms will be measured by patient self-report using the Oral Mucositis Symptom Assessment scale with positive symptoms defined as a score of 1 or greater and severe symptoms defined as a score of 2 or greater.

SECONDARY OUTCOMES:
Incidence and severity of oral mucositis symptoms per chemotherapy cycle | Cycle 1 of chemotherapy (14-28 days, time frame varies based on regimen)
  • The presence and severity of oral mucositis symptoms will be measured by patient self-report using the Oral Mucositis Symptom Assessment scale with positive symptoms defined as a score of 1 or greater and severe symptoms defined as a score of 2 or greater.
Incidence and severity of oral mucositis symptoms per chemotherapy cycle | Cycle 2 of chemotherapy (14-28 days, time frame varies based on regimen)
  • The presence and severity of oral mucositis symptoms will be measured by patient self-report using the Oral Mucositis Symptom Assessment scale with positive symptoms defined as a score of 1 or greater and severe symptoms defined as a score of 2 or greater.
Duration of oral mucositis symptoms | Cycle 1 of chemotherapy (14-28 days, time frame varies based on regimen)
  • The presence and severity of oral mucositis symptoms will be measured by patient self-report using the Oral Mucositis Symptom Assessment scale with positive symptoms defined as a score of 1 or greater and severe symptoms defined as a score of 2 or greater.
Duration of oral mucositis symptoms | Cycle 2 of chemotherapy (14-28 days, time frame varies based on regimen)
  • The presence and severity of oral mucositis symptoms will be measured by patient self-report using the Oral Mucositis Symptom Assessment scale with positive symptoms defined as a score of 1 or greater and severe symptoms defined as a score of 2 or greater.
Percent of days the Chemo MouthpieceTM was used | Cycle 1 of chemotherapy (14-28 days, time frame varies based on regimen)
  • Device use will be measured on a daily diary completed for at least the first 14 days of each cycle. The diary will also be completed on any additional days that the patient uses the device.
Percent of days the Chemo MouthpieceTM was used | Cycle 2 of chemotherapy (14-28 days, time frame varies based on regimen)
  • Device use will be measured on a daily diary completed for at least the first 14 days of each cycle. The diary will also be completed on any additional days that the patient uses the device.
Ease of use of the Chemo MouthpieceTM based on patient-reported Chemo Mouthpiece End of Study Device Assessment | Cycle 1 of chemotherapy (14-28 days, time frame varies based on regimen)
  patient-reported Chemo Mouthpiece End of Study Device Assessment
Ease of use of the Chemo MouthpieceTM based on patient-reported Chemo Mouthpiece End of Study Device Assessment | Cycle 2 of chemotherapy (14-28 days, time frame varies based on regimen)
  patient-reported Chemo Mouthpiece End of Study Device Assessment
Analgesic use to control mouth pain | Cycle 1 of chemotherapy (14-28 days, time frame varies based on regimen)
  Device use will be measured on a daily diary completed for at least the first 14 days of each cycle. The diary will also be completed on any additional days that the patient uses the device.
Analgesic use to control mouth pain | Cycle 2 of chemotherapy (14-28 days, time frame varies based on regimen)
  Device use will be measured on a daily diary completed for at least the first 14 days of each cycle. The diary will also be completed on any additional days that the patient uses the device.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jacobucci, Study Director — Chemo Mouthpiece
Locations (11):
- United States (11):
  - Chan Soon-Shiong Institute for Medicine, Costa Mesa, California
  - Goshen Health, Goshen, Indiana
  - Revive Research Institute, Farmington Hills, Michigan
  - Revive Research Institute, Inc., Sterling Heights, Michigan
  - Phelps Health, Rolla, Missouri
  - Inspira Medical Center, Mullica Hill, New Jersey
  - Inspira Medical Center, Vineland, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - New York Cancer & Blood Specialists, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Gibbs Cancer Center, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zuniga R, Dembla V, Alam N, Nangia C, Guerrero-Garcia T, Chung G, Kio E, Go M, Tubb E, Sonis S, Jacobucci F. Multi-institutional, randomized, controlled trial to assess the efficacy and tolerability of a reusable, self-contained cryotherapy delivery device. Support Care Cancer. 2025 Jul 31;33(8):732. doi: 10.1007/s00520-025-09795-x. PMID 40742459